CLINICAL TRIAL: NCT01041755
Title: The Infusion of L-Ornithine L-aspart is as Effective as Nonabsorbable Disaccharides in the Management of Acute Hepatic Encephalopathy.
Brief Title: Efficacy of L-Ornithine L-Aspartate in Acute Hepatic Encephalopathy.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centro Regional para el Estudio de las Enfermedades Digestivas (Other)
Collaborators: MERZ PHARMA (Unknown)
Responsible Party: Principal Investigator, Dr. Claudia Isabel Blanco Vela, MD, Centro Regional para el Estudio de las Enfermedades Digestivas
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MI09-002
Record Dates: First submitted 2009-12-31; First posted 2010-01-01 (Estimated); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Hepatic Encephalopathy
Keywords: Encephalopathy; Cirrhosis
MeSH Terms: conditions — Hepatic Encephalopathy; Brain Diseases; Fibrosis | interventions — ornithylaspartate; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous infusion of L- Ornithine L- Aspartate (Experimental): a) 20 g L-ornithine-L-aspartate
  Interventions: Drug: L-ornithine-L-aspartate
- Lactose enemas (Active Comparator): b) 20% Lactose enemas
  Interventions: Drug: Lactose

INTERVENTIONS:
Drug: L-ornithine-L-aspartate — a) Intravenous infusion of 20 g L-ornithine-L-aspartate (4 ampules of 10 mL each) in 250 mL sodium chloride solution administered daily in 4 hours for 3 consecutive days, plus the placebo b) Water enemas, 1000 mL of water and given as retention enema every 12 hours for 3 consecutive days.
  Other Names: LOLA
  Arms: Intravenous infusion of L- Ornithine L- Aspartate
Drug: Lactose — a) 20% Lactose enemas, 200 g Lactose diluted with 700 mL of water and given as retention enema every 12 hours for 3 consecutive days, plus intravenous placebo b)250 mL sodium chloride solution, infusion for 4 hours for 3 consecutive days.
  Arms: Lactose enemas

SUMMARY:
Hepatic encephalopathy is caused by the effects on the brain of substances that under normal circumstances are efficiently metabolized in the liver. The hyperammonemia is the main factor responsible for the development of hepatic encephalopathy. In patients with cirrhosis, the reduction in hepatocellular function and generation of portosystemic shunts contribute to increase serum ammonium. The current therapeutic approaches, are aimed at reducing blood ammonium levels.

Administration of the non-absorbable disaccharides, have become standard treatment of hepatic encephalopathy.There are no adequate clinical trials comparing the efficacy of L-Ornithine-L-Aspartate (LOLA) infusion against lactose enemas in the treatment of acute hepatic encephalopathy.

DETAILED DESCRIPTION:
The main impact of hepatic encephalopathy in patients with cirrhosis is not related to costs, but its association with decreased survival and quality of life and should therefore clearly established the effectiveness of therapeutic interventions used in this disorder.

At the end of the nineteenth century to the ammonium was identified as the main agent responsible for the development of the syndrome of hepatic encephalopathy. Since then, reduced nitrogen compounds from the intestine are considered the main therapeutic measure. On this conceptual base, nonabsorbable disaccharides are the first line therapy in hepatic encephalopathy.

Current knowledge indicates that other organs such as muscle, brain and kidney are involved in the generation of ammonium, which has set the pace for the development of new treatments, able to act systemically in metabolism and elimination of ammonia . L-ornithine L-aspartate (LOLA) lowers ammonium concentrations in animal and humans models with hyperammonemia. There are no adequate clinical trials comparing the efficacy of LOLA infusion against lactose enemas in the treatment of acute hepatic encephalopathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cirrhosis of any etiology, diagnosed by ultrasound,clinical and / or histologic criteria
* Patients over 18 years and under 75
* Patients with hepatic encephalopathy grade 3-4 according to the criteria of West Haven
* Patients with hyperammonemia >10 µmol/l

Exclusion Criteria:

* Evidence of neurological or psychiatric illness
* Use of drugs affecting the central nervous system
* Withdrawal Syndrome
* Anorectal disease that interferes with the administration of enemas

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Improvement of at least one grade in mental state based on the West Haven Criteria | 72 hours
  Improvement was assessed at 0, 24, 48 and 72 hours. The mental state was scored from trivial lack of awareness to deep coma from grade 1 to grade 4.

SECONDARY OUTCOMES:
Improvement of at least one grade in mental state assessed by the Glasgow Coma Scale | 72 hours
  Improvement was assessed at 0, 24, 48 and 72 hours. The Glasgow Coma Scale assesses three aspects of responsiveness: eye-opening, motor, and verbal responses. The eye-opening was quantified from 1 to 4 points, the motor response from 1 to 6 points and the verbal response from 1 to 5 points.
Improvement of at least one grade in mental state assessed by the Clinical Hepatic Encephalopathy Staging Scale (CHESS) | 72 hours
  Improvement was assessed at 0, 24, 48 and 72 hours. The CHESS scale has 9 dichotomous questions that assess mental state, intellectual function, behavior, verbal and motor response and orientation. It was quantified from 0 to 9 points.
Improvement of asterixis grade | 72 hours
  Improvement was assessed at 0, 24, 48 and 72 hours. Asterixis was graded as follows: Grade 0 = without flapping motion, Grade 1 ≤ 5 flaps per minute, Grade 2 = 6 to 10 flaps per minute, Grade 3 = 11 to 20 flaps per minute and Grade 4, continuous flap or patient in coma unable to maintain wrist dorsiflexion. Asterixis grade was evaluated at 0. 24, 48 and 72 hours.
Improvement in electroencephalographic tracing grade | 72 hours
  Improvement was assessed at 0 and 72 hours. EEG tracing was graduated from 0 to 4: Grade 0 = normal alpha rhythm, Grade 1 =7 to 8 cycles per second, Grade 2= 5 to 6 cycles per second, Grade 3 = 3 to 4.5 cycles per second and Grade 4 < than 3 cycles per second or delta rhythm. EEG was assessed at 0 and 72 hours.
Improvement in serum ammonia | 72 hours
  Ammonia determination was performed at 0, 24, 48 and 72 hours.
Improvement in Number connection tests | 72 hours
  The mental state of the patients included in the study did not allow them to perform the number connection test, therefore, they were all assigned to the worst score (Grade 4)
Improvement in Portosystemic Encephalopathy Index. | 72 hours
  Improvement was assessed at 0 and 72 hours. The PSE Index was calculated by multiplying the grade of mental state by a factor of 3; and the grades of asterixis, number connection tests, serum ammonia and EEG were multiplied times a factor of 1. The results were divided by the maximal possible PSE sum.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco J Bosques, MD, PhD, Study Director — Centro Regional para el Estudio de las Enfermedades Digestivas; Claudia Isabel Blanco Vela, MD, Principal Investigator — Hospital Juárez de México
Locations (1):
- Hospital Universitario "José Eleuterio González", Monterrey, Nuevo León, Mexico